CLINICAL TRIAL: NCT07335588
Title: A Phase 3, Double-blinded, Vehicle-controlled Trial to Investigate the Efficacy and Safety of Twice Daily Delgocitinib Cream in Adult Participants With Lichen Sclerosus During a 12-Week Initial Treatment Period Followed by a 40-Week Continuation Treatment Period
Brief Title: A 52-Week Trial to Investigate the Efficacy and Safety of Delgocitinib Cream in Adult Participants With Lichen Sclerosus
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0133-2395; 2025-524873-17-00 (EU CTIS Number); U1111-1333-1675 (Other: World Health Organization (WHO))
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lichen Sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — delgocitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1: Delgocitinib Cream 20 mg/g (Experimental): Participants will receive delgocitinib cream 20 mg/g twice daily (BID) in both the 12-week initial treatment period and the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib
- Part 1: Delgocitinib Cream 20 mg/g, then Cream Vehicle (Experimental): Participants will receive delgocitinib cream 20 mg/g BID in the 12-week initial treatment period, then cream vehicle BID in the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib; Drug: Cream Vehicle
- Part 1: Delgocitinib Cream 8 mg/g (Experimental): Participants will receive delgocitinib cream 8 mg/g BID in both the 12-week initial treatment period and the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib
- Part 1: Delgocitinib Cream 8 mg/g, then Cream Vehicle (Experimental): Participants will receive delgocitinib cream 8 mg/g BID in the 12-week initial treatment period, then cream vehicle BID in the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib; Drug: Cream Vehicle
- Part 1: Cream Vehicle, then Delgocitinib Cream 20 mg/g (Experimental): Participants will receive cream vehicle BID in the 12-week initial treatment period, then delgocitinib cream 20 mg/g BID in the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib; Drug: Cream Vehicle
- Part 1: Cream Vehicle, then Delgocitinib Cream 8 mg/g (Experimental): Participants will receive cream vehicle BID in the 12-week initial treatment period, then delgocitinib cream 8 mg/g BID in the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib; Drug: Cream Vehicle
- Part 1: Cream Vehicle (Placebo Comparator): Participants will receive cream vehicle BID in both the 12-week initial treatment period and the 40-week continuation treatment period.
  Interventions: Drug: Cream Vehicle
- Part 2: Delgocitinib Cream (Selected Dose) (Experimental): Participants will receive delgocitinib cream, at the selected dose from Part 1, BID in both the 12-week initial treatment period and the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib
- Part 2: Delgocitinib Cream (Selected Dose), then Cream Vehicle (Experimental): Participants will receive delgocitinib cream, at the selected dose from Part 1, BID in the 12-week initial treatment period, then cream vehicle BID in the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib; Drug: Cream Vehicle
- Part 2: Cream Vehicle, then Delgocitinib Cream (Selected Dose) (Experimental): Participants will receive cream vehicle BID in the 12-week initial treatment period, then delgocitinib cream, at the selected dose from Part 1, BID in the 40-week continuation treatment period.
  Interventions: Drug: Delgocitinib; Drug: Cream Vehicle
- Part 2: Cream Vehicle (Placebo Comparator): Participants will receive cream vehicle BID in both the 12-week initial treatment period and the 40-week continuation treatment period.
  Interventions: Drug: Cream Vehicle

INTERVENTIONS:
Drug: Delgocitinib — Participants will receive delgocitinib BID via topical application.
  Arms: Part 1: Cream Vehicle, then Delgocitinib Cream 20 mg/g; Part 1: Cream Vehicle, then Delgocitinib Cream 8 mg/g; Part 1: Delgocitinib Cream 20 mg/g; Part 1: Delgocitinib Cream 20 mg/g, then Cream Vehicle; Part 1: Delgocitinib Cream 8 mg/g; Part 1: Delgocitinib Cream 8 mg/g, then Cream Vehicle; Part 2: Cream Vehicle, then Delgocitinib Cream (Selected Dose); Part 2: Delgocitinib Cream (Selected Dose); Part 2: Delgocitinib Cream (Selected Dose), then Cream Vehicle
Drug: Cream Vehicle — Participants will receive cream vehicle BID via topical administration.
  Arms: Part 1: Cream Vehicle; Part 1: Cream Vehicle, then Delgocitinib Cream 20 mg/g; Part 1: Cream Vehicle, then Delgocitinib Cream 8 mg/g; Part 1: Delgocitinib Cream 20 mg/g, then Cream Vehicle; Part 1: Delgocitinib Cream 8 mg/g, then Cream Vehicle; Part 2: Cream Vehicle; Part 2: Cream Vehicle, then Delgocitinib Cream (Selected Dose); Part 2: Delgocitinib Cream (Selected Dose), then Cream Vehicle

SUMMARY:
The main purpose of this trial is to learn if female participants have reduced lichen sclerosus (LS) symptoms after treatment with delgocitinib. The researchers are focusing on female participants because LS is more likely to affect females compared to males.

The trial will be conducted in 2 parts. Part 1 of the trial (including dose selection) will only enroll female participants with LS. The selected dose will then be evaluated in Part 2 of the trial, which will be open to both female and male participants with LS. The selected dose will remain blinded in Part 2. Assessment of efficacy and safety of delgocitinib cream in male participants with LS will be evaluated in a substudy.

For each participant, the trial will last at least 55 weeks and up to 60 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Signed and dated informed consent has been obtained prior to any protocol-related procedures.
2. Age ≥18 years at the time of signing informed consent.
3. Participant is able to comply with clinic visits and trial requirements and procedures, as assessed by the investigator.
4. Female participants or male participants (assigned sex at birth and has not had any gender affirming medical procedures to their genital area) with LS in the anogenital area, regardless of treatment history. The diagnosis must be based on typical clinical features and supported by biopsy. A biopsy must be taken if there is no previous documented biopsy to support the diagnosis.

   Note: Participants who also have LS-affected areas outside the anogenital area are allowed to be enrolled but these areas will not be treated with investigational medicinal product (IMP). Participants with newly diagnosed LS can be included, as well as participants who have progressive LS (including existing architectural changes).
5. Disease severity graded as mild to severe at screening and baseline according to IGA-LS score (ie, an IGA-LS score of ≥2).
6. Female participants: A woman of childbearing potential (WOCBP) must agree to use a highly effective or acceptable form of birth control throughout the trial up until the last application of IMP. Male participants: Contraceptive requirements are not applicable for male participants.

Exclusion Criteria

1. Participants with atypical presentation of LS in the anogenital area where the diagnosis is uncertain, or the suspicion of malignancy exists.
2. Female participants: History of vulvar squamous cell carcinoma (SCC), including precursor lesions (eg, human papillomavirus-independent [HPV-I] vulvar intraepithelial neoplasia [VIN] and high-grade squamous intraepithelial lesion). Male participants: History of penile SCC, including precursor lesions.
3. Female participants only: Participants with any abnormal cytology result at screening following a positive high-risk human papillomavirus (hrHPV) screening test.
4. Active dermatologic or gynecologic conditions that could confound the diagnosis of LS or interfere with assessment of the IMP (eg, urinary incontinence-associated dermatitis, genital lichen planus, and genital psoriasis), as assessed by the investigator.
5. Participants with severe urinary incontinence. Incontinence is considered severe if it occurs on most days and more than a few drops at a time.
6. Female participants: Suspected clinically (or confirmed diagnostically) of having active infection in the anogenital area, including candidiasis, Chlamydia trachomatis, Trichomonas vaginalis, Neisseria gonorrhoeae, Mycoplasma genitalium, bacterial vaginosis, or herpes simplex. Participants who test positive for sexually transmitted disease (STD)/bacterial vaginosis (BV)/anogenital candidiasis during screening can be treated, and if repeat testing is negative, these participants can be enrolled. If treatment is needed, the screening period can be extended to 6 weeks to accommodate the treatment and washout requirements.

   Male participants: Suspected clinically (or confirmed diagnostically) of having active infection in the anogenital area, including candidiasis, Chlamydia trachomatis, Neisseria gonorrhoeae, Mycoplasma genitalium, or herpes simplex. Participants who test positive for STD/anogenital candidiasis during screening can be treated, and if repeat testing is negative, these participants can be enrolled. If treatment is needed, the screening period can be extended to 6 weeks to accommodate the treatment and washout requirements.
7. Clinically significant infection within 4 weeks prior to baseline which, in the opinion of the investigator, may compromise the safety of the participant in the trial, interfere with evaluation of the IMP, or reduce the participant's ability to participate in the trial.

   Clinically significant infections are defined as:
   * A systemic infection.
   * A serious skin infection requiring parenteral (intravenous or intramuscular) antibiotics, antiviral, or antifungal medication.
8. History of any known primary immunodeficiency disorder including a positive human immunodeficiency virus test at screening, or the participant taking antiretroviral medications as determined by medical history and/or participant's verbal report.
9. Major surgery within 8 weeks prior to screening or planned in-patient surgery or hospitalization during the trial period.
10. History of cancer:

    • Female participants: Participants who have had basal cell carcinoma or localized SCC of the skin (outside the anogenital area), or in situ carcinoma of the cervix are eligible provided that curative therapy was successfully completed at least 12 months prior to screening.

    Participants who have had other malignancies (except vulvar SCC) are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to screening.

    • Male participants: Participants who have had basal cell carcinoma or localized SCC of the skin (outside the anogenital area) are eligible provided that curative therapy was successfully completed at least 12 months prior to screening.

    Participants who have had other malignancies (except penile SCC) are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to screening.
11. Positive hepatitis B surface antigen and/or hepatitis B core antibody and positive for hepatitis B virus deoxyribonucleic acid (participants who have tested positive for hepatitis B core antibody are eligible if tests for hepatitis B surface antigen and hepatitis B virus deoxyribonucleic acid are negative), or positive hepatitis C virus antibody serology confirmed by hepatitis C virus ribonucleic acid (RNA) at screening.
12. Known or suspected hypersensitivity to any component(s) of the IMP(s).
13. Any disorder which is not stable and according to the investigator could:

    * Affect the safety of the participant throughout the trial.
    * Hinder the participant's ability to complete the trial.

    Examples include, but are not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, immunological, and psychiatric disorders, and major physical impairment.
14. Any abnormal finding which according to the investigator may:

    * Put the participant at risk because of their participation in the trial.
    * Influence the participant's ability to complete the trial.

    The abnormal finding must be clinically significant and observed during the screening period. Examples include abnormal findings in physical examination, vital signs, electrocardiogram (ECG), hematology, or biochemistry.
15. Current or recent chronic alcohol or drug abuse, or any other condition associated with poor compliance as judged by the investigator.
16. Female participants only: Women who are pregnant or lactating. For women of childbearing potential, a negative pregnancy test is required at screening.
17. Systemic treatment with immunosuppressive drugs (eg, methotrexate, cyclosporine), immunomodulating drugs, retinoids, or corticosteroids within 4 weeks prior to baseline.
18. Cutaneously applied treatment with immunomodulators (eg, topical calcineurin inhibitor [TCI]) or topical corticosteroid (TCS) on the anogenital area within 2 weeks before baseline.
19. Use of systemic or topical Janus kinase (JAK) inhibitors (including delgocitinib) within 4 weeks before baseline.
20. Systemic or cutaneous (applied in the anogenital area) use of antibiotics, antiparasitics, antivirals, or antifungals within 1 week before baseline.
21. Treatment with any marketed biological therapy or investigational biologic agents:

    * Any cell-depleting agent including but not limited to rituximab: within 6 months prior to baseline, or until the lymphocyte count returns to normal, whichever is longer.
    * Other biologics: within 3 months or 5 half-lives, whichever is longer, prior to baseline.
22. Treatment with any non-marketed drug substance (that is, an agent that has not yet been made available for clinical use following registration) within 4 weeks prior to baseline or 5 half-lives, whichever is longer.
23. Light-based therapy on the anogenital area and treatments with platelet-rich plasma within 4 weeks prior to baseline.
24. Cutaneous treatments applied within 1 week before baseline in regions other than the anogenital area which could interfere with clinical trial evaluations or pose a safety concern.
25. Other cutaneous therapies or therapeutic procedures on the anogenital area within 1 week before baseline.
26. Surgical treatment for anogenital LS in the past 6 months or have not recovered fully from an earlier surgical procedure in the anogenital area.
27. Female participants only: Participants who are receiving doses that are not stable for topical estrogens (<4 weeks before screening), and hormonal contraceptives and hormone replacement therapy (HRT) medications (<3 months before screening).
28. Current participation in any other interventional clinical trial.
29. Previously randomized in this clinical trial.
30. Previously randomized in a clinical trial with delgocitinib.
31. Clinically important laboratory abnormalities:

    * Participants with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values ≥2×the upper limit of normal (ULN) with total bilirubin (BIL) ≥1.5×ULN (unless elevated BIL is related to Gilbert Meulengracht Syndrome).
    * Participants with ALT and/or AST values ≥3×ULN.
    * Participants with severe renal impairment (estimated glomerular filtration rate [eGFR]<30 mL/min/1.73 m2).
32. Employees of the trial site, or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals.
33. Participants who are legally institutionalized.
34. Only applicable in France: Participant not affiliated with or not a beneficiary of a social security scheme.
35. Male participants only: Participants who currently need or are expected during the entire study period to require any type of surgical treatment for LS (eg, circumcision, urethroplasty, adhesiolysis) or tool-assisted local treatment (eg, catheter, cotton swabs, applicators, dilators, etc.) for LS involving the urethra. Application of study treatment of the urethral meatus is allowed if it can be applied by the participant's hand or fingers only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2026-05-06 (Estimated); Primary Completion 2028-03-10 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving IGA-LS TS at Week 12 | Week 12

SECONDARY OUTCOMES:
Number of Participants Achieving IGA-LS TS at Week 8 | Week 8
Change in Clinical Lichen Sclerosus Score (CLISSCO) from Baseline to Week 12 | Baseline to Week 12
Number of Participants Achieving a Reduction of Skin Pain Numerical Rating Scale (NRS) Score (Weekly Average) of ≥4 Points from Baseline to Week 12 in Participants with Baseline Skin Pain NRS Score ≥4 | Baseline to Week 12
Number of Participants Achieving a Reduction of Skin Pain NRS Score (Weekly Average) of ≥4 Points from Baseline to Week 8 in Participants with Baseline Skin Pain NRS Score ≥4 | Baseline to Week 8
Number of Participants Achieving a Reduction of Itch NRS Score (Weekly Average) of ≥4 Points from Baseline to Week 12 in Participants with Baseline Itch NRS Score ≥4 | Baseline to Week 12
Number of Participants Achieving a Reduction of Itch NRS Score (Weekly Average) of ≥4 Points from Baseline to Week 8 in Participants with Baseline Itch NRS Score ≥4 | Baseline to Week 8
Change in Vulvar Quality of Life Index (VQLI) Score from Baseline to Week 12 | Baseline to Week 12
Number of Participants Achieving IGA-LS TS at Week 52 | Week 52
Change in CLISSCO Score from Baseline to Week 52 | Baseline to Week 52
Number of Participants Achieving IGA-LS TS at Week 52 Among Participants Having Achieved IGA-LS TS at Week 12 | Week 52
Number of Participants Achieving an IGA-LS Score of 0 or 1 at Week 52 Among Participants Having Achieved IGA-LS TS at Week 12 | Week 52
Time to IGA-LS TS from Baseline to Week 52 | Baseline to Week 52
Time to IGA-LS ≥2 from Week 12 to Week 52 Among Participants Having Achieved IGA-LS TS at Week 12 | Week 12 to Week 52
Number of Participants Having no Increase in CLISSCO Architectural Changes Domain Score from Baseline to Week 52 | Baseline to Week 52
Number of Participants Achieving a Reduction of Skin Pain NRS Score (Weekly Average) of ≥4 Points from Baseline to Week 52 in Participants with Baseline Skin Pain NRS Score ≥4 | Baseline to Week 52
Number of Participants Achieving a Reduction of Itch NRS Score (Weekly Average) of ≥4 Points from Baseline to Week 52 in Participants with Baseline Itch NRS Score ≥4 | Baseline to Week 52
Number of Treatment-emergent Adverse Events (TEAEs) from Baseline to Week 12 | Baseline to Week 12
Number of TEAEs from Week 12 to Week 54 | Week 12 to Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma

IPD SHARING:
Plan to Share IPD: No